CLINICAL TRIAL: NCT01314261
Title: A Blinded, Randomized, Placebo-Controlled, Dose-Ranging Study to Evaluate the Safety, Pharmacokinetics, and Antiviral Activity of ABT-267 in Combination With Peginterferon Alpha-2a and Ribavirin (pegIFN/RBV) in Treatment-Naïve Subjects With Genotype 1 Chronic Hepatitis C Virus (HCV) Infection
Brief Title: Study of ABT-267 in Treatment Naive Hepatitis C Virus (HCV) Genotype 1 Infected Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M12-114
Record Dates: First submitted 2011-03-11; First posted 2011-03-14 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2015-01

CONDITIONS: Chronic Hepatitis C; Hepatitis C Virus (HCV) Infection
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C; Infections | interventions — ombitasvir; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- ABT-267 (5 mg) once daily + pegIFN/RBV (Experimental): Participants were given 5 mg ABT-267 once daily in combination with pegylated interferon/ribavirin (pegIFN/RBV) for 12 weeks, followed by 36 weeks of pegIFN/RBV treatment alone. Pegylated interferon was dosed 180 µg subcutaneously once a week. Ribavirin was dosed 1000 or 1200 mg daily divided twice a day.
  Interventions: Drug: ABT-267; Drug: Pegylated interferon (pegIFN); Drug: Ribavirin (RBV)
- ABT-267 (50 mg) once daily + pegIFN/RBV (Experimental): Participants were given 50 mg ABT-267 once daily in combination with pegylated interferon/ribavirin (pegIFN/RBV) for 12 weeks, followed by 36 weeks of pegIFN/RBV treatment alone. Pegylated interferon was dosed 180 µg subcutaneously once a week. Ribavirin was dosed 1000 or 1200 mg daily divided twice a day.
  Interventions: Drug: ABT-267; Drug: Pegylated interferon (pegIFN); Drug: Ribavirin (RBV)
- ABT-267 (200 mg) once daily + pegIFN/RBV (Experimental): Participants were given 200 mg ABT-267 once daily in combination with pegylated interferon/ribavirin (pegIFN/RBV) for 12 weeks, followed by 36 weeks of pegIFN/RBV treatment alone. Pegylated interferon was dosed 180 µg subcutaneously once a week. Ribavirin was dosed 1000 or 1200 mg daily divided twice a day.
  Interventions: Drug: ABT-267; Drug: Pegylated interferon (pegIFN); Drug: Ribavirin (RBV)
- Placebo + pegIFN/RBV (Placebo Comparator): Participants were given matching placebo to ABT-267 once daily in combination with pegIFN/RBV for 12 weeks, followed by 36 weeks of pegIFN/RBV treatment alone. Pegylated interferon was dosed 180 µg subcutaneously once a week. Ribavirin was dosed 1000 or 1200 mg daily divided twice a day.
  Interventions: Drug: Pegylated interferon (pegIFN); Drug: Ribavirin (RBV); Other: Placebo for ABT-267

INTERVENTIONS:
Drug: ABT-267 — 5 mg or 25 mg tablets
  Other Names: Ombitasvir
  Arms: ABT-267 (200 mg) once daily + pegIFN/RBV; ABT-267 (5 mg) once daily + pegIFN/RBV; ABT-267 (50 mg) once daily + pegIFN/RBV
Drug: Pegylated interferon (pegIFN) — Syringe, 180 µg/0.5 mL for subcutaneous injections administered weekly
Drug: Ribavirin (RBV) — 200 mg tablet dosed at 1000 or 1200 mg daily divided twice a day
Other: Placebo for ABT-267 — Participants received matching placebo tablet at each dose level for ABT-267.
  Arms: Placebo + pegIFN/RBV

SUMMARY:
The purpose of this study was to assess the safety, pharmacokinetics, and 4-week rapid virologic response (RVR) of 3 different doses of ABT-267 (also known as ombitasvir) in combination with pegylated interferon/ribavirin (pegIFN/RBV) compared with pegIFN/RBV alone (ABT-267 placebo) in treatment naïve, hepatitis C virus (HCV), genotype 1-infected participants.

DETAILED DESCRIPTION:
The study was a randomized, double blind, placebo controlled study consisting of 2 substudies. In substudy 1, participants received 1 of 3 doses of ABT-267 or placebo + pegIFN/RBV for 12 weeks. In substudy 2, participants received pegIFN/RBV for 36 weeks. Participants were followed for 48 weeks post ABT-267 treatment for evaluation of efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Treatment naïve participants
* Females must be either postmenopausal for at least 2 years or surgically sterile
* Males must be surgically sterile or practicing specific forms of birth control
* Chronic hepatitis C virus (HCV), genotype-1 infected participants
* Documented FibroTest score in combination with an Aspartate Aminotransferase to Platelet Ratio Index (APRI), or a liver biopsy within the last 12 months to document absence of cirrhosis

Exclusion Criteria:

* Pregnant or breastfeeding female
* Use of any medications contraindicated for use with pegylated interferon(pegIFN) or ribavirin (RBV) 2 weeks prior to study drug administration or 10 half-lives, whichever is longer
* Clinically significant cardiac, respiratory (except mild asthma), renal, gastrointestinal, hematologic, neurologic disease, or any uncontrolled medical illness or psychiatric disease or disorder
* Current or past clinical evidence of cirrhosis or bridging fibrosis
* Abnormal screening laboratory results

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-03; Primary Completion 2012-01 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Armen Asatryan, MD, Study Director — AbbVie
Locations (11):
- United States (10):
  - Site Reference ID/Investigator# 56623, Birmingham, Alabama
  - Site Reference ID/Investigator# 48476, Los Angeles, California
  - Site Reference ID/Investigator# 51345, Orlando, Florida
  - Site Reference ID/Investigator# 51498, Honolulu, Hawaii
  - Site Reference ID/Investigator# 48473, Indianapolis, Indiana
  - Site Reference ID/Investigator# 52782, Kansas City, Missouri
  - Site Reference ID/Investigator# 48471, Houston, Texas
  - Site Reference ID/Investigator# 48474, San Antonio, Texas
  - Site Reference ID/Investigator# 48477, Fairfax, Virginia
  - Site Reference ID/Investigator# 48472, Seattle, Washington
- Site Reference ID/Investigator# 48483, San Juan, Puerto Rico

REFERENCES:
- [Background] Mensing S, Polepally AR, Konig D, Khatri A, Liu W, Podsadecki TJ, Awni WM, Menon RM, Dutta S. Population Pharmacokinetics of Paritaprevir, Ombitasvir, Dasabuvir, Ritonavir, and Ribavirin in Patients with Hepatitis C Virus Genotype 1 Infection: Combined Analysis from 9 Phase 1b/2 Studies. AAPS J. 2016 Jan;18(1):270-80. doi: 10.1208/s12248-015-9846-1. Epub 2015 Nov 23. PMID 26597291
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ABT-267 (5 mg) Once Daily + pegIFN/RBV | ABT-267 (50 mg) Once Daily + pegIFN/RBV | ABT-267 (200 mg) Once Daily + pegIFN/RBV | Placebo + pegIFN/RBV
Started | 9 | 9 | 10 | 9
Discontinued ABT-267 or Placebo | 1 | 0 | 1 | 0
Discontinued pegIFN/RBV | 1 | 4 | 5 | 1
Completed | 7 | 5 | 7 | 6
Not Completed | 2 | 4 | 3 | 3
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 2 | 2
Not completed — Virologic Failure | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All 37 participants enrolled in the study received at least 1 dose of study drug and were included in the intent-to-treat population for efficacy and safety analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | ABT-267 (5 mg) Once Daily + pegIFN/RBV | ABT-267 (50 mg) Once Daily + pegIFN/RBV | ABT-267 (200 mg) Once Daily + pegIFN/RBV | Placebo + pegIFN/RBV | Total
Number analyzed (Participants) | 9 | 9 | 10 | 9 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (11.32) | 49.2 (9.55) | 46.0 (10.26) | 48.1 (12.32) | 48.3 (10.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 4 | 4 | 15
  Male | 4 | 7 | 6 | 5 | 22

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With 4-week Rapid Virologic Response (RVR)
Description: Plasma hepatitis C virus ribonucleic acid (HCV RNA) levels (measured in IU/mL) were determined for each sample using a real-time reverse transcriptase-polymerase chain reaction (RT-PCR) assay. Rapid virologic response was defined as HCV RNA levels < the lower limit of detection (< 15 IU/mL) at Week 4. Data are reported as percentage of participants with RVR.
Time Frame: Week 4
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | ABT-267 (5 mg) Once Daily + pegIFN/RBV | ABT-267 (50 mg) Once Daily + pegIFN/RBV | ABT-267 (200 mg) Once Daily + pegIFN/RBV | Placebo + pegIFN/RBV
Number analyzed (Participants) | 9 | 9 | 10 | 9
percentage of participants | 33.3 | 55.6 | 70.0 | 22.2
Statistical Analysis 1: Comparison: ABT-267 (5 mg) Once Daily + pegIFN/RBV vs Placebo + pegIFN/RBV; Ten participants in an ABT-267 arm and nine participants in the placebo arm would provide 84% power using Fisher's exact test with two-sided significance level of 0.05 to detect a difference of approximately 70% between the two arms; Test type: Superiority or Other; p = 0.336, Regression, Logistic — No adjustments were made for multiple comparisons and the pre-specified, two-sided significance level was 0.05; Treatment group, baseline HCV RNA level, HCV subgenotype (1a or 1b), and interleukin 28B genotype (CC or non-CC) were predictors
Statistical Analysis 2: Comparison: ABT-267 (50 mg) Once Daily + pegIFN/RBV vs Placebo + pegIFN/RBV; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.171, Regression, Logistic — No adjustments were made for multiple comparisons and the pre-specified, two-sided significance level was 0.05; Treatment group, baseline HCV RNA level, HCV sub-genotype (1a or 1b), and interleukin 28B genotype (CC or non-CC) were predictors
Statistical Analysis 3: Comparison: ABT-267 (200 mg) Once Daily + pegIFN/RBV vs Placebo + pegIFN/RBV; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.030, Regression, Logistic — No adjustments were made for multiple comparisons and the pre-specified, two-sided significance level was 0.05; [statistical method as in outcome 1, analysis 2]

2. Secondary Outcome: Percentage of Participants With Partial Early Virologic Response (pEVR)
Description: Plasma hepatitis C virus ribonucleic acid (HCV RNA) levels (measured in IU/mL) were determined for each sample using a real-time reverse transcriptase-polymerase chain reaction (RT-PCR) assay. Partial EVR was defined as HCV RNA levels that decreased > 2 log10 IU/mL at Week 12 as compared to baseline HCV RNA levels. Data are reported as the percentage of participants with pEVR.
Time Frame: Baseline and Week 12
Population: All 37 participants enrolled in the study received at least 1 dose of study drug and were included in the intent-to-treat population for efficacy analyses.
Measure: Number; unit: percentage of participants
Arm/Group | ABT-267 (5 mg) Once Daily + pegIFN/RBV | ABT-267 (50 mg) Once Daily + pegIFN/RBV | ABT-267 (200 mg) Once Daily + pegIFN/RBV | Placebo + pegIFN/RBV
Number analyzed (Participants) | 9 | 9 | 10 | 9
percentage of participants | 100.0 | 88.9 | 90.0 | 77.8
Statistical Analysis 1: Comparison: ABT-267 (5 mg) Once Daily + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.102, Cochran-Mantel-Haenszel — No adjustments were made for multiple comparisons and the pre-specified, two-sided significance level was 0.05; Controlled for interleukin 28B genotype (CC or non-CC), HCV sub-genotype (1a or 1b), and baseline HCV RNA levels (≤ median or > median)
Statistical Analysis 2: Comparison: ABT-267 (50 mg) Once Daily + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.362, Cochran-Mantel-Haenszel — No adjustments were made for multiple comparisons and the pre-specified, two-sided significance level was 0.05; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: ABT-267 (200 mg) Once Daily + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.079, Cochran-Mantel-Haenszel — No adjustments were made for multiple comparisons and the pre-specified, two-sided significance level was 0.05; [statistical method as in outcome 2, analysis 1]

3. Primary Outcome: Maximum Plasma Concentration (Cmax) of ABT-267
Description: Blood samples were collected immediately prior to morning dose (time 0 hours); 2, 4, 6, and 8 hours after the morning dose on Day 1; and prior to dose on Day 2 (24 hours after Day 1 dose). The samples were analyzed for the concentration of ABT-267 using validated analytical methods. The maximum plasma concentration (Cmax; measured in ng/mL) is the highest concentration that a drug achieves in the plasma after administration in a dosing interval. The Cmax of ABT-267 was estimated using non-compartmental methods and data are reported as the mean ± standard deviation.
Time Frame: Immediately prior to morning dose (time 0 hours); 2, 4, 6, and 8 hours after the morning dose on Day 1; and prior to dose on Day 2 (24 hours after Day 1 dose)
Population: Participants received at least 1 dose of study drug and had sufficient concentrations to characterize the pharmacokinetic parameters.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ABT-267 (5 mg) Once Daily + pegIFN/RBV | ABT-267 (50 mg) Once Daily + pegIFN/RBV | ABT-267 (200 mg) Once Daily + pegIFN/RBV
Number analyzed (Participants) | 9 | 9 | 9
ng/mL | 10.7 (3.73) | 148 (80.8) | 535 (160)

4. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) of ABT-267
Description: Blood samples were collected immediately prior to morning dose (time 0 hours); 2, 4, 6, and 8 hours after the morning dose on Day 1; and prior to dose on Day 2 (24 hours after Day 1 dose). The samples were analyzed for the concentration of ABT-267 using validated analytical methods. The time to maximum plasma concentration (Tmax; measured in hours) is the time it takes for a drug to achieve Cmax. The Tmax of ABT-267 was estimated using non-compartmental methods and data are reported as the mean ± standard deviation.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | ABT-267 (5 mg) Once Daily + pegIFN/RBV | ABT-267 (50 mg) Once Daily + pegIFN/RBV | ABT-267 (200 mg) Once Daily + pegIFN/RBV
Number analyzed (Participants) | 9 | 9 | 9
Hours | 3.3 (1.0) | 3.8 (1.6) | 4.2 (1.6)

5. Primary Outcome: Area Under the Plasma Concentration-time Curve From 0 to 24 Hours (AUC24) Post-dose of ABT-267
Description: Blood samples were collected immediately prior to morning dose (time 0 hours); 2, 4, 6, and 8 hours after the morning dose on Day 1; prior to dose on Day 2 (24 hours after Day 1 dose); and at each subsequent study visit. The samples were analyzed for the concentration of ABT-267 using validated analytical methods. The area under the plasma concentration -time curve (AUC; measured in ng*hr/mL) is a method of measurement of the total exposure of a drug in blood plasma. The AUC24 of ABT-267 was estimated using non-compartmental methods and data are reported as the mean ± standard deviation.
Time Frame: Immediately prior to morning dose (time 0 hours); 2, 4, 6, and 8 hours after the morning dose on Day 1; prior to dose on Day 2 (24 hours after Day 1 dose); and at each subsequent study visit up to Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | ABT-267 (5 mg) Once Daily + pegIFN/RBV | ABT-267 (50 mg) Once Daily + pegIFN/RBV | ABT-267 (200 mg) Once Daily + pegIFN/RBV
Number analyzed (Participants) | 7 | 3 | 4
ng*hr/mL | 115 (35.5) | 2200 (1090) | 6130 (675)

6. Secondary Outcome: Percentage of Participants With Complete Early Virologic Response (cEVR)
Description: Plasma hepatitis C virus ribonucleic acid (HCV RNA) levels (measured in IU/mL) were determined for each sample using a real-time reverse transcriptase-polymerase chain reaction (RT-PCR) assay. Complete EVR was defined as HCV RNA < the lower limit of quantification (< 25 IU/mL) at Week 12. Data are reported as the percentage of participants with cEVR.
Time Frame: Week 12
Population: All 37 participants enrolled in the study received at least 1 dose of study drug and were included in the intent-to-treat population for efficacy analysis.
Measure: Number; unit: percentage of participants
Arm/Group | ABT-267 (5 mg) Once Daily + pegIFN/RBV | ABT-267 (50 mg) Once Daily + pegIFN/RBV | ABT-267 (200 mg) Once Daily + pegIFN/RBV | Placebo + pegIFN/RBV
Number analyzed (Participants) | 9 | 9 | 10 | 9
percentage of participants | 100.0 | 88.9 | 80.0 | 66.7
Statistical Analysis 1: Comparison: ABT-267 (5 mg) Once Daily + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.083, Cochran-Mantel-Haenszel — No adjustments were made for multiple comparisons and the pre-specified, two-sided significance level was 0.05; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: ABT-267 (50 mg) Once Daily + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.515, Cochran-Mantel-Haenszel — No adjustments were made for multiple comparisons and the pre-specified, two-sided significance level was 0.05; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: ABT-267 (200 mg) Once Daily + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.221, Cochran-Mantel-Haenszel — No adjustments were made for multiple comparisons and the pre-specified, two-sided significance level was 0.05; [statistical method as in outcome 2, analysis 1]

7. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks (SVR12) Post-pegylated Interferon/Ribavirin (pegIFN/RBV) Dosing
Description: Plasma hepatitis C virus ribonucleic acid (HCV RNA) levels (measured in IU/mL) were determined for each sample using a real-time reverse transcriptase-polymerase chain reaction (RT-PCR) assay. Sustained virologic response was defined as HCV RNA levels < the lower limit of quantification (< 25 IU/mL) 12 weeks after the last dose of pegIFN/RBV. Data are reported as the percentage of participants with SVR12.
Time Frame: 12 weeks after the last dose of pegIFN/RBV
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | ABT-267 (5 mg) Once Daily + pegIFN/RBV | ABT-267 (50 mg) Once Daily + pegIFN/RBV | ABT-267 (200 mg) Once Daily + pegIFN/RBV | Placebo + pegIFN/RBV
Number analyzed (Participants) | 9 | 9 | 10 | 9
percentage of participants | 66.7 | 66.7 | 60.0 | 33.3
Statistical Analysis 1: Comparison: ABT-267 (5 mg) Once Daily + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.155, Regression, Logistic — No adjustments were made for multiple comparisons and the pre-specified, two-sided significance level was 0.05; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: ABT-267 (50 mg) Once Daily + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.214, Regression, Logistic — No adjustments were made for multiple comparisons and the pre-specified, two-sided significance level was 0.05; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: ABT-267 (200 mg) Once Daily + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.231, Regression, Logistic — No adjustments were made for multiple comparisons and the pre-specified, two-sided significance level was 0.05; [statistical method as in outcome 1, analysis 2]

8. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 24 Weeks (SVR24) Post-pegylated Interferon/Ribavirin (pegIFN/RBV) Dosing
Description: Plasma hepatitis C virus ribonucleic acid (HCV RNA) levels (measured in IU/mL) were determined for each sample using a real-time reverse transcriptase-polymerase chain reaction (RT-PCR) assay. Sustained virologic response was defined as HCV RNA levels < the lower limit of quantification (< 25 IU/mL) 24 weeks after the last dose of pegIFN/RBV. Data are reported as the percentage of participants with SVR24.
Time Frame: 24 weeks after the last dose of pegIFN/RBV
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | ABT-267 (5 mg) Once Daily + pegIFN/RBV | ABT-267 (50 mg) Once Daily + pegIFN/RBV | ABT-267 (200 mg) Once Daily + pegIFN/RBV | Placebo + pegIFN/RBV
Number analyzed (Participants) | 9 | 9 | 10 | 9
percentage of participants | 55.6 | 44.4 | 50.0 | 22.2
Statistical Analysis 1: Comparison: ABT-267 (5 mg) Once Daily + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.127, Regression, Logistic — No adjustments were made for multiple comparisons and the pre-specified, two-sided significance level was 0.05; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: ABT-267 (50 mg) Once Daily + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.328, Regression, Logistic — No adjustments were made for multiple comparisons and the pre-specified, two-sided significance level was 0.05; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: ABT-267 (200 mg) Once Daily + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.166, Regression, Logistic — No adjustments were made for multiple comparisons and the pre-specified, two-sided significance level was 0.05; [statistical method as in outcome 1, analysis 2]

9. Secondary Outcome: Median Time to Suppression of Hepatitis C Virus Ribonucleic Acid (HCV RNA)
Description: Plasma hepatitis C virus ribonucleic acid (HCV RNA) levels (measured in IU/mL) were determined for each sample using a real-time reverse transcriptase-polymerase chain reaction (RT-PCR) assay. Time to suppression was defined as the time (measured in days) to HCV RNA levels < the lower limit of quantification (< 25 IU/mL). Data are reported as the median number of days.
Time Frame: Approximately 12 weeks
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | ABT-267 (5 mg) Once Daily + pegIFN/RBV | ABT-267 (50 mg) Once Daily + pegIFN/RBV | ABT-267 (200 mg) Once Daily + pegIFN/RBV | Placebo + pegIFN/RBV
Number analyzed (Participants) | 9 | 9 | 10 | 9
Days | 27.0 [7.0 to 43.0] | 16.0 [7.0 to 42.0] | 21.5 [7.0 to 29.0] | 84.0 [NA to NA] — The confidence limit for the placebo group is not calculated as the participants were either suppressed at Week 12 (end of the time frame), or never suppressed and censored at Week 12.
Statistical Analysis 1: Comparison: ABT-267 (5 mg) Once Daily + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.007, Log Rank — No adjustments were made for multiple comparisons and the pre-specified, two-sided significance level was 0.05
Statistical Analysis 2: Comparison: ABT-267 (50 mg) Once Daily + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.029, Log Rank — No adjustments were made for multiple comparisons and the pre-specified, two-sided significance level was 0.05
Statistical Analysis 3: Comparison: ABT-267 (200 mg) Once Daily + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.105, Log Rank — No adjustments were made for multiple comparisons and the pre-specified, two-sided significance level was 0.05

10. Primary Outcome: Plasma Concentrations of Ribavirin (RBV)
Description: Blood samples were collected at each study visit from Week 1 to Week 12. The samples were analyzed for the concentration of RBV (measured in ng/mL) using validated analytical methods and RBV concentrations in plasma were summarized at each visit. Data are reported as the median (range).
Time Frame: At each study visit from Week 1 to Week 12
Population: Participants received at least 1 dose of study drug and had sufficient concentrations to characterize the pharmacokinetic parameters. When a different number of participants at a specific time point was used to analyze the data in the outcome measure, the n (number of participants) for each arm is denoted in the Category Title.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | ABT-267 (5 mg) Once Daily + pegIFN/RBV | ABT-267 (50 mg) Once Daily + pegIFN/RBV | ABT-267 (200 mg) Once Daily + pegIFN/RBV | Placebo + pegIFN/RBV
Number analyzed (Participants) | 9 | 9 | 10 | 9
ng/mL
  Week 1 | 1330 [852 to 3950] | 1470 [847 to 2700] | 1060 [742 to 1700] | 1190 [860 to 2130]
  Week 2 | 1890 [484 to 6160] | 1640 [328 to 3810] | 1420 [1140 to 2150] | 1360 [1130 to 2740]
  Week 4 (n=8, 8, 10, 9) | 1900 [1110 to 4500] | 1680 [279 to 3290] | 1580 [1250 to 2110] | 1950 [842 to 3520]
  Week 6 (n=8, 9, 9, 9) | 2000 [1390 to 3250] | 1510 [0.00 to 3210] | 1780 [890 to 2280] | 1900 [1380 to 4300]
  Week 8 (n=8, 9, 9, 9) | 2080 [712 to 3400] | 1710 [277 to 3160] | 1650 [1120 to 2290] | 2280 [277 to 4630]
  Week 12 (n=8, 9, 9, 9) | 2510 [1300 to 4320] | 1740 [0.00 to 2240] | 1800 [1270 to 2590] | 1940 [0.00 to 4760]

11. Primary Outcome: Serum Concentrations of Pegylated Interferon (pegIFN)
Description: Blood samples were collected at each study visit from Week 1 to Week 12. The samples were analyzed for the concentration of pegIFN (measured in ng/mL) using validated analytical methods and pegIFN concentrations in serum were summarized at each visit. Data are reported as the median (range).
Time Frame: At each study visit from Week 1 to Week 12
Population: as for outcome 10
Measure: Median (Full Range); unit: ng/mL
Arm/Group | ABT-267 (5 mg) Once Daily + pegIFN/RBV | ABT-267 (50 mg) Once Daily + pegIFN/RBV | ABT-267 (200 mg) Once Daily + pegIFN/RBV | Placebo + pegIFN/RBV
Number analyzed (Participants) | 9 | 9 | 10 | 9
ng/mL
  Week 1 | 7.50 [2.08 to 13.4] | 6.12 [2.26 to 9.83] | 4.30 [0.00 to 13.9] | 4.83 [2.09 to 20.0]
  Week 2 | 8.75 [4.00 to 24.4] | 9.22 [4.64 to 14.4] | 7.52 [0.00 to 20.1] | 6.87 [1.04 to 16.4]
  Week 4 (n=9, 9, 10, 9) | 11.8 [2.97 to 26.2] | 7.72 [3.07 to 16.1] | 8.23 [0.00 to 23.4] | 8.76 [5.12 to 16.9]
  Week 6 (n=8, 9, 9, 9) | 10.9 [6.09 to 21.0] | 9.35 [5.20 to 15.9] | 14.6 [3.59 to 24.1] | 10.9 [6.21 to 17.3]
  Week 8 (n=8, 9, 9, 9) | 9.91 [5.40 to 22.7] | 10.1 [2.47 to 15.7] | 12.1 [3.94 to 30.3] | 11.0 [4.74 to 17.8]
  Week 12 (n=8, 9, 9, 9) | 14.4 [4.83 to 24.2] | 6.16 [0.00 to 15.3] | 15.2 [6.39 to 25.6] | 8.91 [0.00 to 19.3]

12. Secondary Outcome: Percentage of Participants With Extended Rapid Virologic Response (eRVR)
Description: Plasma hepatitis C virus ribonucleic acid (HCV RNA) levels (measured in IU/mL) were determined for each sample using a real-time reverse transcriptase-polymerase chain reaction (RT-PCR) assay. Extended RVR was defined as HCV RNA levels < the lower level of quantification (< 25 IU/mL) at Weeks 4 through 12. Data are reported as the percentage of participants with eRVR.
Time Frame: Week 4 through Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | ABT-267 (5 mg) Once Daily + pegIFN/RBV | ABT-267 (50 mg) Once Daily + pegIFN/RBV | ABT-267 (200 mg) Once Daily + pegIFN/RBV | Placebo + pegIFN/RBV
Number analyzed (Participants) | 9 | 9 | 10 | 9
percentage of participants | 77.8 | 77.8 | 80.0 | 22.2
Statistical Analysis 1: Comparison: ABT-267 (5 mg) Once Daily + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.028, Regression, Logistic — No adjustments were made for multiple comparisons and the pre-specified, two-sided significance level was 0.05; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: ABT-267 (50 mg) Once Daily + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.051, Regression, Logistic — No adjustments were made for multiple comparisons and the pre-specified, two-sided significance level was 0.05; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: ABT-267 (200 mg) Once Daily + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.021, Regression, Logistic — No adjustments were made for multiple comparisons and the pre-specified, two-sided significance level was 0.05; [statistical method as in outcome 1, analysis 2]

ADVERSE EVENTS:
Time Frame: Non-serious adverse events were collected from the time of study drug administration to 30 days after last dose of study drug (ABT-267 or placebo; 16 Weeks).
Description: A treatment-emergent adverse event was defined as any event with an onset date that was after the first dose of ABT-267/placebo and no more than 30 days after the last dose of ABT-267 or placebo.
Groups:
- ABT-267 (5 mg) Once Daily + pegIFN/RBV: Participants were given 5 mg ABT-267 once daily in combination with pegylated interferon/ribavirin (pegIFN/RBV) for 12 weeks. Pegylated interferon was dosed 180 µg subcutaneously once a week. Ribavirin was dosed 1000 or 1200 mg daily divided twice a day.
- ABT-267 (50 mg) Once Daily + pegIFN/RBV: Participants were given 10 mg ABT-267 once daily in combination with pegylated interferon/ribavirin (pegIFN/RBV) for 12 weeks. Pegylated interferon was dosed 180 µg subcutaneously once a week. Ribavirin was dosed 1000 or 1200 mg daily divided twice a day.
- ABT-267 (200 mg) Once Daily + pegIFN/RBV: Participants were given 200 mg ABT-267 once daily in combination with pegylated interferon/ribavirin (pegIFN/RBV) for 12 weeks. Pegylated interferon was dosed 180 µg subcutaneously once a week. Ribavirin was dosed 1000 or 1200 mg daily divided twice a day.
- Placebo + pegIFN/RBV: Participants were given matching placebo to ABT-267 once daily in combination with pegIFN/RBV for 12 weeks. Pegylated interferon was dosed 180 µg subcutaneously once a week. Ribavirin was dosed 1000 or 1200 mg daily divided twice a day.
Arm/Group | ABT-267 (5 mg) Once Daily + pegIFN/RBV | ABT-267 (50 mg) Once Daily + pegIFN/RBV | ABT-267 (200 mg) Once Daily + pegIFN/RBV | Placebo + pegIFN/RBV
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 9/9 | 9/9 | 8/10 | 9/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABT-267 (5 mg) Once Daily + pegIFN/RBV (N=9) | ABT-267 (50 mg) Once Daily + pegIFN/RBV (N=9) | ABT-267 (200 mg) Once Daily + pegIFN/RBV (N=10) | Placebo + pegIFN/RBV (N=9)
ANAEMIA (Blood and lymphatic system disorders) | 2 | 2 | 2 | 0
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 2 | 1 | 2 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
PALPITATIONS (Cardiac disorders) | 0 | 1 | 0 | 0
EAR DISCOMFORT (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
VERTIGO (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
BLEPHARITIS (Eye disorders) | 0 | 0 | 1 | 0
EYE INFLAMMATION (Eye disorders) | 0 | 1 | 0 | 0
VISION BLURRED (Eye disorders) | 0 | 1 | 0 | 0
VISUAL IMPAIRMENT (Eye disorders) | 0 | 0 | 1 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 0 | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 1 | 0
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 | 0 | 0 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 0 | 1 | 1
ABDOMINAL TENDERNESS (Gastrointestinal disorders) | 0 | 0 | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 2 | 1 | 1 | 1
DRY MOUTH (Gastrointestinal disorders) | 0 | 0 | 1 | 0
FLATULENCE (Gastrointestinal disorders) | 0 | 0 | 1 | 0
GLOSSITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 1
NAUSEA (Gastrointestinal disorders) | 2 | 3 | 4 | 3
STOMATITIS (Gastrointestinal disorders) | 0 | 1 | 0 | 0
TONGUE DISORDER (Gastrointestinal disorders) | 0 | 0 | 1 | 0
TOOTHACHE (Gastrointestinal disorders) | 0 | 0 | 1 | 1
VOMITING (Gastrointestinal disorders) | 2 | 2 | 3 | 2
CHILLS (General disorders) | 3 | 2 | 1 | 0
FATIGUE (General disorders) | 7 | 6 | 5 | 6
FEELING ABNORMAL (General disorders) | 0 | 1 | 0 | 0
GAIT DISTURBANCE (General disorders) | 0 | 1 | 0 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 0 | 1 | 0 | 2
INJECTION SITE ERYTHEMA (General disorders) | 1 | 0 | 2 | 1
IRRITABILITY (General disorders) | 1 | 0 | 0 | 1
NODULE (General disorders) | 0 | 0 | 1 | 0
PAIN (General disorders) | 3 | 1 | 3 | 0
PYREXIA (General disorders) | 1 | 1 | 1 | 0
ABSCESS LIMB (Infections and infestations) | 0 | 0 | 1 | 0
BRONCHITIS (Infections and infestations) | 1 | 1 | 0 | 1
ORAL FUNGAL INFECTION (Infections and infestations) | 0 | 1 | 0 | 0
SINUSITIS (Infections and infestations) | 1 | 0 | 0 | 0
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 | 0 | 1 | 0
TOOTH ABSCESS (Infections and infestations) | 0 | 0 | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0 | 0
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
LACERATION (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
BLOOD GLUCOSE INCREASED (Investigations) | 0 | 0 | 1 | 0
WEIGHT DECREASED (Investigations) | 0 | 1 | 1 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 | 2 | 1 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
DISTURBANCE IN ATTENTION (Nervous system disorders) | 0 | 1 | 0 | 0
DIZZINESS (Nervous system disorders) | 1 | 1 | 0 | 0
HEADACHE (Nervous system disorders) | 3 | 3 | 3 | 2
HYPERAESTHESIA (Nervous system disorders) | 0 | 1 | 0 | 0
MEMORY IMPAIRMENT (Nervous system disorders) | 0 | 1 | 0 | 0
MIGRAINE (Nervous system disorders) | 0 | 0 | 1 | 0
PSYCHOMOTOR HYPERACTIVITY (Nervous system disorders) | 0 | 0 | 1 | 0
TREMOR (Nervous system disorders) | 0 | 0 | 0 | 1
ANXIETY (Psychiatric disorders) | 0 | 2 | 2 | 2
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 0 | 1 | 1
DEPRESSION (Psychiatric disorders) | 1 | 1 | 2 | 1
INSOMNIA (Psychiatric disorders) | 2 | 1 | 1 | 2
MOOD ALTERED (Psychiatric disorders) | 0 | 0 | 1 | 0
MOOD SWINGS (Psychiatric disorders) | 0 | 0 | 1 | 0
NIGHTMARE (Psychiatric disorders) | 0 | 0 | 1 | 0
RESTLESSNESS (Psychiatric disorders) | 0 | 0 | 1 | 0
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
POSTMENOPAUSAL HAEMORRHAGE (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
DRY SKIN (Skin and subcutaneous tissue disorders) | 3 | 1 | 1 | 1
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
HEAT RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 3 | 0 | 3 | 2
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
RASH GENERALISED (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
URTICARIA (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
HOT FLUSH (Vascular disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.